CLINICAL TRIAL: NCT06638606
Title: Microbiota Profiles in Newly Married Couples: Potential Effects on Vision, Sleep and Psychometric Parameters
Status: Enrolling by invitation | Type: Observational
Sponsor: Reza Rastmanesh (Other)
Responsible Party: Sponsor-Investigator, Reza Rastmanesh, Principal Investigator, Shahid Beheshti University of Medical Sciences
Organization: Shahid Beheshti University of Medical Sciences (Other)
Other Study IDs: it24412; it24412 (Other: National Science Institute, Iran); IT. 24001670 (Other: National Science Foundation, Iran)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Sleep Deprivation; Gut Microbiota; Optometry Examinations; Oral Microbiota; Depression; Anxiety
Keywords: Depression; Anxiety; Oral microbiota; Saliva cortisol
MeSH Terms: conditions — Sleep Deprivation; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Oral, fecal and conjunctival samples will be collected from participants and will be stored (at - 20, and - 80◦C, respectively) until further processing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A: Normal couples (have normal sleep pattern), B: Insomniac and C: hypersomniac couples: Group A: Couples with normal sleep pattern. Group B: One spouse suffers from insomnia. Group C: Once spouse suffers from hypersomnia.
  Interventions: Behavioral: Sleep improvement techniques

INTERVENTIONS:
Behavioral: Sleep improvement techniques — Insomniac and hypersomniac individuals are given behavioral counselling to improve sleep.

SUMMARY:
Oral, fecal and conjunctival samples will be collected from participants and will be stored (at - 20 and - 80 ◦C) until further processing. On Day 1 and Day 2, all couples will participate in an oral, conjunctival and gut microbiota composition study. Optometry examinations will be completed for each participant Three and Six months later, oral, conjunctival and gut microbiota composition will be analyzed again with the same protocol. The participants will complete a validated Persian version of Pittsburgh Sleep Quality Inventory (PSQI), Epworth Sleepiness Scale (ESS), Insomnia Severity Index (ISI), global sleep assessment questionnaire (GSAQ) and Ocular Surface Disease Index.

Consecutive couples will undergo a standard ophthalmology exam and specific assessments for dry eye, including non-anesthetic Schirmer's test and fluorescein tear break-up time on Day 1 and Day 90.

DETAILED DESCRIPTION:
The metabolic activity, diversity and composition of the gut microbiota vary significantly between healthy individuals and insomniacs, and also between hypersomniacs and healthy people. While Clostridiales and Bacteroides are regarded to be the two most important biomarkers for differentiating between healthy people and insomniacs, a recent study demonstrated that an enhanced relative abundance of five genera including Lachnospiraceae UCG010, Hungatella, Collinsella, Gordonibacter and Blautia may be correlated with a diminished risk of some types of hypersomnia (narcolepsy type one). Contrarily, an enhanced relative abundance of class Betaproteobacteria, genus Ruminiclostridium and genus Alloprevotella may potentially increase the risk of narcolepsy type one.

Furthermore, recent studies demonstrated that there were no significant differences in alpha and beta diversity between the three groups nonmyopes (NM), progressive myopes (progressive myopes ) and stable myopes (SM). Nothwithstanding, the distributions of Dorea, Roseburia,, Faecalibacterium, Coprococcus, Bacteroides, Bifidobacterium, Megamonas, and Blautia were significantly higher in the myopes (SM and PM combined) when compared with emmetropes. The myopes showed significantly higher abundance of bacteria that are linked to the regulation of dopaminergic signalling, such as Bacteroides, Ruminococcus, Clostridium, Bifidobacterium. Participants with stable myopia were found to have a significantly higher proportion of Prevotella copri than those with progressive myopia. Bifidobacterium adolescentis, a gamma-aminobutyric acid (GABA)-producing bacterium, was significantly higher in all myopes than in NM and, in the comparison between SM and PM, it is significantly higher in SM. B. uniformis and B. fragilis, both GABA-producing Bacteroides, were present in relatively high abundance in all myopes and in SM compared with PM, respectively.

Some researches have detected substantial bacterial strain sharing across people with distinct intra-population, mother-to-infant and intra-household transmission patterns. There was considerable strain sharing among cohabiting people, with 32% and 12% median strain-sharing rates for the time since cohabitation and gut and oral microbiomes affected strain sharing more than genetics or age did.

Salivary samples were collected from all participant. Couples were instructed not to consume any food or drink, except water, for at least 30 min prior to sample collection. Saliva cortisol was then measured by LC-MS/MS as described before.

The validated Persian version Beck Depression Inventory-II (BDI-II), Beck Anxiety Inventory (BAI), and Pittsburgh Sleep Quality Index (PSQI) will be employed to measure depression, anxiety, and sleep quality, respectively.

Insomnia in this study is defined as coexistence of both daytime dysfunction and difficulty resuming sleep. Hypersomnia is defined by a bed-rest total sleep time ≥19 hours during the 32-hour recording. SPSS software will be used to analyze the data.

Based on these premises, below hypotheses are proposed:

* Person-to-person bacterial transmission can change the sleep pattern in newly married couples through gut microbiota
* Person-to-person bacterial transmission can alter vision status in newly married couples through ocular microbiota
* Person-to-person bacterial transmission can alter depression and anxiety status in newly married couples through ocular microbiota

ELIGIBILITY:
Inclusion Criteria:

* Sleep disorder (insomnia and hypersomnia)
* Depressive/anxiety states

Exclusion Criteria:

* Medicines known to affect gut/oral/ocular microbiota composition
* Pregnant/pregnancy
* Divorce during the study
* Antibiotics use in the past month
* Ongoing, active ocular infection, including conjunctivitis.
* Not having any prior history with Dry eye disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All volunteer participants who had been officially married during the past six months and are in a cohabiting relationship will be invited to participate in this study together with their official spouses.
Sampling Method: Non-Probability Sample
Enrollment: 1740 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Sleep Pattern | 3 months later, sleep quality and quantity will be measured with Pittsburgh Sleep Quality Inventory
  Sleep quality and quantity will be evaluated using Pittsburgh Sleep Quality Inventory.
Optometry examinations | 3 months
Depression | 6 months later, will be measured using Beck Anxiety Inventory-II.
  The BDI-II is a commonly utilized 21-item self-report inventory designed for assessing depressive symptomatology, referring to the last two weeks. Higher scores demonstrate more severe depressive symptomatology. Depression in this study was defined as a BDI-II score ≥14
Anxiety | 6 months later, will be measured using Beck Anxiety Inventory
  BAI questionnaire has 21 items with scores ranging from 0-3 for each item, in which 0 indicates "not at all," 1 indicates "mildly, but it did not bother me much," 2 indicates "moderately, it was not pleasant at times," and 3 indicates "severely, it bothered me a lot" for all the items.

SECONDARY OUTCOMES:
Dry eye symptom | at 3, 6 and 12 months will be measured using Ocular Surface Disease Index (OSDI) questionnaire
  Dry eye disease (DED) will be evaluated using Ocular Surface Disease Index questionnaire. DED is classified as mild (13-22 points), moderate (23-32 points), or severe (33-100 points).

CONTACTS AND LOCATIONS:
Overall Officials: Reza Rastmanesh Principal investigator, unaffilaited, PhD, Principal Investigator; Abolfazl Sadeghinejad, MD, Study Director; Javid Azizi, MD, Study Director
Locations (1):
- Private sleep clinic, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
Oral, fecal and conjunctival samples will be collected from participants and will be stored according to the standard protocols until further processing. On Day 1 and Day 2, all couples will participate in a gut microbiota composition study. Optometry examinations will be completed for each participant Three months later, gut microbiota composition will be analyzed again with the same protocol. The participants will complete a validated Persian version of Pittsburgh Sleep Quality Inventory (PSQI), Epworth Sleepiness Scale (ESS), Insomnia Severity Index (ISI), and global sleep assessment questionnaire (GSAQ). Insomnia in this study is defined as coexistence of both daytime dysfunction and difficulty resuming sleep. Hypersomnia is defined by a bed-rest total sleep time ≥19 hours during the 32-hour recording. SPSS software will be used to analyze the data.
  For more detail, contact me: r.rastmanesh@gmail.com

REFERENCES:
- [Background] Zhang J, Lu X, Cheng Z, Zou D, Shi W, Wang T. Alterations of conjunctival microbiota associated with orthokeratology lens wearing in myopic children. BMC Microbiol. 2023 Dec 13;23(1):397. doi: 10.1186/s12866-023-03042-1. PMID 38087200
- [Background] Omar WEW, Singh G, McBain AJ, Cruickshank F, Radhakrishnan H. Gut Microbiota Profiles in Myopes and Nonmyopes. Invest Ophthalmol Vis Sci. 2024 May 1;65(5):2. doi: 10.1167/iovs.65.5.2. PMID 38691091
- [Background] Wu Y, Fan H, Feng Y, Yang J, Cen X, Li W. Unveiling the gut microbiota and metabolite profiles in guinea pigs with form deprivation myopia through 16S rRNA gene sequencing and untargeted metabolomics. Heliyon. 2024 May 6;10(9):e30491. doi: 10.1016/j.heliyon.2024.e30491. eCollection 2024 May 15. PMID 38756593
- [Background] Zhang Y, Zhou X, Lu Y. Gut microbiota and derived metabolomic profiling in glaucoma with progressive neurodegeneration. Front Cell Infect Microbiol. 2022 Aug 12;12:968992. doi: 10.3389/fcimb.2022.968992. eCollection 2022. PMID 36034713
- [Background] Li H, Liu S, Zhang K, Zhu X, Dai J, Lu Y. Gut microbiome and plasma metabolome alterations in myopic mice. Front Microbiol. 2023 Dec 21;14:1251243. doi: 10.3389/fmicb.2023.1251243. eCollection 2023. PMID 38179454
- [Background] Sun Y, Xie Y, Li J, Hou X, Sha Y, Bai S, Yu H, Liu Y, Wang G. Study on the relationship between adolescent myopia and gut microbiota via 16S rRNA sequencing. Exp Eye Res. 2024 Oct;247:110067. doi: 10.1016/j.exer.2024.110067. Epub 2024 Sep 3. PMID 39233303
- [Background] Li H, Du Y, Cheng K, Chen Y, Wei L, Pei Y, Wang X, Wang L, Zhang Y, Hu X, Lu Y, Zhu X. Gut microbiota-derived indole-3-acetic acid suppresses high myopia progression by promoting type I collagen synthesis. Cell Discov. 2024 Aug 27;10(1):89. doi: 10.1038/s41421-024-00709-5. PMID 39187483
- [Background] Walters EM, Phillips AJ, Hamill K, Norton PJ, Drummond SP. Anxiety predicts dyadic sleep characteristics in couples experiencing insomnia but not in couples without sleep disorders. J Affect Disord. 2020 Aug 1;273:122-130. doi: 10.1016/j.jad.2020.04.031. Epub 2020 May 12. PMID 32421592
- [Background] Saini EK, Keiley MK, Fuller-Rowell TE, Duke AM, El-Sheikh M. Socioeconomic Status and Sleep among Couples. Behav Sleep Med. 2021 Mar-Apr;19(2):159-177. doi: 10.1080/15402002.2020.1721501. Epub 2020 Feb 2. PMID 32008377
- [Background] Gunn HE, Buysse DJ, Hasler BP, Begley A, Troxel WM. Sleep Concordance in Couples is Associated with Relationship Characteristics. Sleep. 2015 Jun 1;38(6):933-9. doi: 10.5665/sleep.4744. PMID 25581920
- [Background] Coutinho J, Pereira A, Oliveira-Silva P, Meier D, Lourenco V, Tschacher W. When our hearts beat together: Cardiac synchrony as an entry point to understand dyadic co-regulation in couples. Psychophysiology. 2021 Mar;58(3):e13739. doi: 10.1111/psyp.13739. Epub 2020 Dec 23. PMID 33355941
- [Background] Liu S, Rovine MJ, Klein LC, Almeida DM. Synchrony of diurnal cortisol pattern in couples. J Fam Psychol. 2013 Aug;27(4):579-88. doi: 10.1037/a0033735. PMID 23978320
- [Background] Evangelista E, Lopez R, Barateau L, Chenini S, Bosco A, Jaussent I, Dauvilliers Y. Alternative diagnostic criteria for idiopathic hypersomnia: A 32-hour protocol. Ann Neurol. 2018 Feb;83(2):235-247. doi: 10.1002/ana.25141. Epub 2018 Feb 9. PMID 29323727
- [Background] Itani O, Kaneita Y, Munezawa T, Mishima K, Jike M, Nakagome S, Tokiya M, Ohida T. Nationwide epidemiological study of insomnia in Japan. Sleep Med. 2016 Sep;25:130-138. doi: 10.1016/j.sleep.2016.05.013. Epub 2016 Aug 30. PMID 27823706
- [Background] Chehri A, Goldaste N, Ahmadi S, Khazaie H, Jalali A. Psychometric properties of insomnia severity index in Iranian adolescents. Sleep Sci. 2021 Apr-Jun;14(2):101-106. doi: 10.5935/1984-0063.20200045. PMID 34381573
- [Background] Valles-Colomer M, Blanco-Miguez A, Manghi P, Asnicar F, Dubois L, Golzato D, Armanini F, Cumbo F, Huang KD, Manara S, Masetti G, Pinto F, Piperni E, Puncochar M, Ricci L, Zolfo M, Farrant O, Goncalves A, Selma-Royo M, Binetti AG, Becerra JE, Han B, Lusingu J, Amuasi J, Amoroso L, Visconti A, Steves CM, Falchi M, Filosi M, Tett A, Last A, Xu Q, Qin N, Qin H, May J, Eibach D, Corrias MV, Ponzoni M, Pasolli E, Spector TD, Domenici E, Collado MC, Segata N. The person-to-person transmission landscape of the gut and oral microbiomes. Nature. 2023 Feb;614(7946):125-135. doi: 10.1038/s41586-022-05620-1. Epub 2023 Jan 18. PMID 36653448
- [Background] Sheng D, Li P, Xiao Z, Li X, Liu J, Xiao B, Liu W, Zhou L. Identification of bidirectional causal links between gut microbiota and narcolepsy type 1 using Mendelian randomization. Sleep. 2024 Mar 11;47(3):zsae004. doi: 10.1093/sleep/zsae004. PMID 38174762
- [Background] Rakoff-Nahoum S, Foster KR, Comstock LE. The evolution of cooperation within the gut microbiota. Nature. 2016 May 12;533(7602):255-9. doi: 10.1038/nature17626. Epub 2016 Apr 25. PMID 27111508
- [Background] Busch A, Roy S, Helbing DL, Colic L, Opel N, Besteher B, Walter M, Bauer M, Refisch A. Gut microbiome in atypical depression. J Affect Disord. 2024 Mar 15;349:277-285. doi: 10.1016/j.jad.2024.01.060. Epub 2024 Jan 9. PMID 38211751
- [Background] Jezkova J, Sonka K, Kreisinger J, Prochazkova P, Tlaskalova-Hogenova H, Nevsimalova S, Buskova J, Merkova R, Dvorakova T, Prihodova I, Dostalova S, Roubalova R. Guardians of Rest? Investigating the gut microbiota in central hypersomnolence disorders. Sleep Med. 2024 Jan;113:95-102. doi: 10.1016/j.sleep.2023.11.024. Epub 2023 Nov 19. PMID 37995475
- [Background] Han M, Yuan S, Zhang J. The interplay between sleep and gut microbiota. Brain Res Bull. 2022 Mar;180:131-146. doi: 10.1016/j.brainresbull.2021.12.016. Epub 2022 Jan 13. PMID 35032622
- [Background] Wang Z, Wang Z, Lu T, Chen W, Yan W, Yuan K, Shi L, Liu X, Zhou X, Shi J, Vitiello MV, Han Y, Lu L. The microbiota-gut-brain axis in sleep disorders. Sleep Med Rev. 2022 Oct;65:101691. doi: 10.1016/j.smrv.2022.101691. Epub 2022 Aug 31. PMID 36099873